CLINICAL TRIAL: NCT05042297
Title: Combined Posterior and Anterior Ring Fixation Versus Posterior Ring Fixation Alone in Management of Unstable Tile B2 and C1 Pelvic Ring Injuries: A Randomized Controlled Trial
Brief Title: Combined Ring (APR) Fixation Vs Posterior Ring Fixation in Tile B2 and C1 Pelvic Ring Injuries
Acronym: APR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Islam Moussa, Assistant lecturer of orthopedic surgery, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD 272/2019
Record Dates: First submitted 2021-09-01; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Evaluation of PR Fixation in Tile B2 and C1 Injuries
Keywords: Tile B2 and C1 pelvic ring injuries; Posterior ring fixation; Sacroiliac Screw; Radiological outcome; Majeed Pelvic Score

STUDY DESIGN:
Intervention Model Description: An independent doctor created the randomization sequence using Excel 2016 (computerized random numbers) with a 1:1 allocation via random block sizes of 2, 4, and 6; he assigned the sample numbers equally to each group and assigned the block. Patients and physicians allocated to each intervention group were aware of the allocation; however, the data analysts and the outcome assessors were kept blinded to the allocation. We prospectively carried out this study on 40 patients with Tile B2 & C1 injuries between March 2019 and July 2020 that met our inclusion criteria. The independent doctor allocated the 40 cases to two groups: Group A (20 cases): combined posterior and anterior ring fixation (APR fixation group), group B (20 cases): isolated posterior ring fixation (PR fixation group).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Patients and physicians allocated to each intervention group were aware of the allocation; however, the data analysts and the outcome assessors were kept blinded to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Posterior and anterior ring fixation (Active Comparator): Posterior ring fixation via a single posterior Sacroiliac screw or two Iliac wing plates. While anterior ring fixation was via a single para-symphyseal plate in Tile B2 injuries. Meanwhile, we used double superior and anterior symphyseal plates in Tile C1 injuries.
  Interventions: Procedure: Combined posterior and anterior ring fixation: Active comparator. Isolated posterior ring fixation: Experimental intervention
- Isolated Posterior ring fixation (Experimental): We used either two Sacroiliac screws in S1 and S2, or two Iliac wing plates.
  Interventions: Procedure: Combined posterior and anterior ring fixation: Active comparator. Isolated posterior ring fixation: Experimental intervention

INTERVENTIONS:
Procedure: Combined posterior and anterior ring fixation: Active comparator. Isolated posterior ring fixation: Experimental intervention — Reduction of the posterior ring was either closed reduction in SI joint dislocations & fracture-dislocations and sacral fractures or open reduction in iliac wing fractures through the lateral window of the ilioinguinal approach. Anterior pelvic ring reduction and fixation in the combined APR fixation group was done via the classic Pfannenstiel approach or extension more lateral & completing the anterior intrapelvic approach. Fixation was via pubic rami plating.

SUMMARY:
The aim for surgical treatment of unstable Tile B2 & C1 pelvic ring injuries is an anatomical reduction to allow early weight-bearing, pain relief and to prevent future pelvic asymmetry. So, we usually used combined posterior & anterior ring fixation, relying on the fact that anterior pelvic ring adequate reduction and fixation better augment posterior ring fixation and enhance overall pelvic stability. However, anterior ring fixation requires a second incision with a longer operation time and more blood loss. The main disadvantage of the second incision is the higher risk of wound infection, either superficial or deep, which questions its necessity and raises concerns about the possibility of isolated posterior ring fixation in managing Tile B2 & C1 pelvic ring injuries with good outcomes.

The fundamental algorithm was the questionable need for additional anterior ring fixation in managing Tile B2 and C1 pelvic ring injuries combined with posterior ring fixation, whether the incidence of postoperative complications, radiological and clinical outcomes differed between these two groups. After reviewing the literature, we found a lack of knowledge in the prospective assessment of such outcomes between the two fixation groups. So, This RCT aims to reach a satisfactory result and prove or deny the questionable need for anterior ring fixation in managing Tile B2 and C1 pelvic ring injuries. Our hypothesis was that PR fixation is at least as good as APR fixation.

DETAILED DESCRIPTION:
Type of Study: Prospective randomized controlled clinical trial Randomization technique: Block Randomization. Study Setting: The operations were held in Ain Shams university hospitals. Study Period: From 2019 till 2020.

Study Population:

Inclusion Criteria:

Tile B2 and C1 pelvic ring injuries Nakatani zone II pubic rami fractures with intact inguinal ligament Age between 16-60 years old Recent pelvic ring injuries less than three weeks

Exclusion Criteria:

Tile A pelvic ring injuries Nakatani zone I & III pubic rami fractures neglected pelvic ring injuries exceeding three weeks Age less than 16 years and older than 60 years

Sampling Method: convenient sample. Sample Size: 40 feet subdivided randomly via Block Randomization into 2 groups, 20 feet for each group.

Group A: Patients treated by combined posterior and anterior ring fixation Group B: Patients treated by posterior ring fixation alone

Ethical Considerations: were followed by obtaining the hospital Research Ethics Committee approval and written informed consents from the patients.

Study Tools:

The patients were evaluated by the following: -

All patients were subjected to:

I. Pre-operative:

Written consent.

Complete ATLS protocol:

Primary survey: airway, breathing, circulation and disability with complete exposure, including: CXR and pelvis anteroposterior view Secondary survey: head to toe examination, complete cervical clinical and radiological clearance and detailed AMPLE history

Detailed history:

History-taking included age, mode of trauma, physiological status, haemodynamics, associated internal organ injuries, medical comorbidities and detailed surgical history.

Complete Orthopaedic examination:

Full and thorough examination of the patient was done from head to toes with complete inspection, palpation and range of motion examination of the whole body, together with detailed neurovascular examination of both lower limbs.

X-Rays pre and post-operative Preoperative: to assess the fracture pattern, location and for surgical planning.

Postoperatively: to assess the quality of reduction immediate postoperative and at each follow up visit (two weeks, six weeks, three months, six months and one year) to follow up union rate, fixation failure, secondary dislocation and secondary loss of reduction.

CT pelvis preoperative will be done to accurately describe fracture pattern, identify occult radiological instability and more comprehensive surgical planning.

Evaluation of the patients by clinical Majeed pelvic scoring system

II.Operative technique Group A: combined posterior and anterior ring fixation Group B: Isolated Posterior ring fixation

III. Postoperative management and evaluation:

We followed a partially assisted weight-bearing protocol for six weeks for both groups (using axillary or forearm crutches that take about 50% of the body weight through the injured lower extremity). In addition, we did x-ray films & neurovascular examination postoperatively.

Follow-up visits were at two weeks, six weeks, three months, six months & 1-year postoperative.

We performed radiological and clinical assessments: Radiological using Matta & Tornetta radiological principles via plain x-ray pelvis showing both hips: anteroposterior, inlet and outlet views & CT pelvis if available; we evaluated five criteria on X-ray films postoperatively: residual posterior displacement, vertical displacement, pubic symphyseal translation, sagittal rotation, and gapping of the sacroiliac joint; according to the grading of Matta and Tornetta, we classified the results into Excellent (less than or equal 4 mm), Good (4-10 mm), Fair (10-20 mm), and Poor (more than 20 mm). In addition, clinical assessment by Majeed pelvic scoring system evaluated and calculated at each follow-up visit with the mean value presented, Postoperative complications and need for another operation were evaluated.

In week two, we encouraged passive and active-assisted hip ROM. Then we started an unassisted weight-bearing and physiotherapy program to strengthen abductors and quadriceps muscles in week six. While complete full weight-bearing and return to work were after three months. After six months, a full radiological and clinical assessment were done + return to pre-injury mobility status and athletic sports. Finally, after one year, we did clinical and radiological reevaluation.

IV- Statistical analysis of data.

V- Outcome measures of interest:

Primary outcomes: radiological (using Matta & Tornetta radiological principles) & clinical outcomes (using the Majeed pelvic scoring system), and postoperative complications.

Secondary outcomes: operative time, amount of blood loss, intraoperative assessment of reduction, need for another operation, length of hospital stay, ability to weight bear postoperative, and pain control metrics.

ELIGIBILITY:
Inclusion Criteria:

* Tile B2 and C1 pelvic ring injuries
* Nakatani zone II pubic rami fractures with intact inguinal ligament
* Age between 16-60 years old
* recent pelvic ring injuries less than three weeks

Exclusion Criteria:

* Tile A pelvic ring injuries
* Nakatani zone I & III pubic rami fractures
* neglected pelvic ring injuries exceeding three weeks
* Age less than 16 years and older than 60 years

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-09 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Rate of Excellent, Good, Fair, or Poor Radiological Outcomes | one year postoperative
  Radiological assessment using Matta & Tornetta radiological principles via plain x-ray pelvis showing both hips: anteroposterior, inlet and outlet views & CT pelvis if available; we evaluated five criteria on X-ray films postoperatively: residual posterior displacement, vertical displacement, pubic symphyseal translation, sagittal rotation, and gapping of the sacroiliac joint; according to the grading of Matta and Tornetta, we classified the results into Excellent (less than or equal 4 mm), Good (4-10 mm), Fair (10-20 mm), and Poor (more than 20 mm).
Rate of Excellent, Good, or Fair Clinical Outcomes | one year postoperative
  clinical assessment by Majeed pelvic scoring system evaluated and calculated at each follow-up visit with the mean value presented
Postoperative Complications' Rate | Through study completion, an average of 1 year postoperative
  We focused the evaluation of Postoperative complications on the local complications related to fixation principles and technique rather than general complications related to the patient status and associated injuries: LLD, foot drop, SI screw cut out, wound infection, residual malunion or non-union of the anterior or posterior ring, and loss of reduction (2ry SI dislocation or any rotational or vertical re-displacement that exceeds 2 cm or posterior sacral fracture gap that exceeds 1 cm)

SECONDARY OUTCOMES:
Mean Operative Time | It was calculated intra-operative
  The mean operation time was calculated and compared between the two study groups
Mean Intraoperative Blood Loss | Up to 4 days postoperative
  The mean blood loss was calculated and compared between the two study groups, it was measured intraoperative and postoperative from suction drains
Need For Another Operations' Rate | Through study completion, an average of 1 year postoperative
  The need for another operation was observed and compared between the two study groups
Rate of Anatomical, Acceptable, or Non-anatomic Intraoperative Assessment of Reduction | It was performed intraoperative
  The intraoperative assessment of reduction was performed and compared the results between the two study groups
The Average Length OF Hospital Stay | Up to 4 days postoperative
  The average hospital stay postoperative was calculated and compared between the two study groups
Number of participants Able To Weight-bear Postoperative | Up to one year postoperative
  We observed the ability of the patients to toe-touch weight-bear immediate postoperative, and it was compared between the two study groups
Number of participants that required IV Opiods as an Analgesia | up to 4 days postoperative
  The analgesica requirements between the two study groups were analyzed and compared, it ranged from users of paracetamol to those who needed IV opiods

CONTACTS AND LOCATIONS:
Overall Officials: Amr K. Mahmoud, Professor, Principal Investigator — no funding recieved
Locations (1):
- Ain Shams University, Cairo, Abassia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmal H, Froberg L, S Larsen M, Sudkamp NP, Pohlemann T, Aghayev E, Goodwin Burri K. Evaluation of strategies for the treatment of type B and C pelvic fractures: results from the German Pelvic Injury Register. Bone Joint J. 2018 Jul;100-B(7):973-983. doi: 10.1302/0301-620X.100B7.BJJ-2017-1377.R1. PMID 29954203
- [Result] Pohlemann T, Stengel D, Tosounidis G, Reilmann H, Stuby F, Stockle U, Seekamp A, Schmal H, Thannheimer A, Holmenschlager F, Gansslen A, Rommens PM, Fuchs T, Baumgartel F, Marintschev I, Krischak G, Wunder S, Tscherne H, Culemann U. Survival trends and predictors of mortality in severe pelvic trauma: estimates from the German Pelvic Trauma Registry Initiative. Injury. 2011 Oct;42(10):997-1002. doi: 10.1016/j.injury.2011.03.053. Epub 2011 Apr 22. PMID 21513936
- [Result] Hauschild O, Strohm PC, Culemann U, Pohlemann T, Suedkamp NP, Koestler W, Schmal H. Mortality in patients with pelvic fractures: results from the German pelvic injury register. J Trauma. 2008 Feb;64(2):449-55. doi: 10.1097/TA.0b013e31815982b1. PMID 18301214
- [Result] Osterhoff G, Ossendorf C, Wanner GA, Simmen HP, Werner CM. Percutaneous iliosacral screw fixation in S1 and S2 for posterior pelvic ring injuries: technique and perioperative complications. Arch Orthop Trauma Surg. 2011 Jun;131(6):809-13. doi: 10.1007/s00402-010-1230-0. Epub 2010 Dec 28. PMID 21188399
- [Result] Sagi HC, Coniglione FM, Stanford JH. Examination under anesthetic for occult pelvic ring instability. J Orthop Trauma. 2011 Sep;25(9):529-36. doi: 10.1097/BOT.0b013e31822b02ae. PMID 21857421